CLINICAL TRIAL: NCT06929286
Title: COMparative Prospective Assessment Through Clinically Integrated Randomized Trials Evaluating Intravesical Treatments: The COMPARE IT Trial
Brief Title: A Study Comparing Standard Treatments in People With Non-Muscle Invasive Bladder Cancer (NMIBC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-069
Record Dates: First submitted 2025-04-14; First posted 2025-04-16 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Non-Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nadofaragene firadenovec (Experimental): The patient will receive nadofaragene firadenovec.
  Interventions: Drug: Nadofaragene Firadenovec
- Best usual care (Active Comparator): For patients randomized to receive best usual care, the combination of intravesical GemDoce is the current standard of care at MSK for most patients with BCG failure.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Nadofaragene Firadenovec — For patients randomized to receive nadofaragene firadenovec, the patient will receive nadofaragene firadenovec as of normal saline instilled intravesically every 3 months for up to 12 months.
  Arms: Nadofaragene firadenovec
Drug: Gemcitabine — gemcitabine instilled intravesically for 1 h, then drained completely out of the bladder
  Arms: Best usual care
Drug: Docetaxel — followed by docetaxel instilled intravesically for 1 h. This is given once weekly for 6 weeks for induction. Those who have a complete response typically proceed with once-monthly instillations of GemDoce for up to 24 months as maintenance therapy
  Arms: Best usual care

SUMMARY:
The purpose of this study is to compare the effectiveness of different FDA-approved/NCCN-recommended drug treatments for NMIBC. In particular, the FDA-approved drug nadofaragene firadenovec will be compared to usual care with other NCCN-recommended standard treatments for NMIBC (gemcitabine with or without docetaxel, mitomycin, re-treatment with BCG, or pembrolizumab).

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Being treated for high-grade NMIBC (Tis, Ta, or T1) with one of the participating treating urologists at MSK
* One or more prior induction course of BCG at any point in time and judgment by the treating urologist that BCG has failed

  °Any amount of maintenance BCG is allowed
* In the previous 12 months, receipt of at least one instillation of any intravesical agent (induction or maintenance) or one administration of systemic therapy for NMIBC treatment

  °An intravesical agent can include BCG or any other NMIBC treatment
* In the opinion of the treating urologist, there is no contraindication to treatment with nadofaragene firadenovec (i.e. hypersensitivity to IFNa, severe immunosuppression) and there is uncertainty over whether nadofaragene is better than "best usual care"

Exclusion Criteria:

* Opting for treatment with radical cystectomy
* Currently enrolled in a clinical trial of an experimental therapy for NMIBC
* Prior exposure to nadofaragene firadenovec

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
high-grade recurrence-free survival | up to 24 months
  The time from the initiation of treatment to the detection of recurrence of high-grade bladder cancer (biopsy-proven intravesical recurrence or distant metastasis). Biopsy proven high grade intravesical recurrence will be based on the MSK pathology review of the bladder tissue samples.

SECONDARY OUTCOMES:
Progression-free survival | up to 24 months
  Disease progression is defined as the development of muscle-invasive disease (stage ≥T2), lymph node or distant metastasis, or death without documented disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Pietzak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm